CLINICAL TRIAL: NCT03923543
Title: Is Neutrophil to Lymphocyte Ratio a Prognostic Factor of Sepsis in Newborns With Operated Congenital Heart Disease
Status: Completed | Type: Observational
Sponsor: Firat Ergin (Other)
Responsible Party: Sponsor-Investigator, Firat Ergin, Dr. Fırat ERGİN, Tepecik Training and Research Hospital
Organization: Tepecik Training and Research Hospital (Other)
Other Study IDs: (2018/12- 7
Record Dates: First submitted 2019-04-17; First posted 2019-04-22 (Actual); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Sepsis Newborn
MeSH Terms: conditions — Neonatal Sepsis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Neutrophil to lymphosit ratio

SUMMARY:
The use of neutrophil lymphocyte ratio is useful for the detection of infection status in newborns after surgery

DETAILED DESCRIPTION:
The use of neutrophil lymphocyte ratio is useful for the detection of infection status in newborns after surgery and we compare this with other acute phase reactants

ELIGIBILITY:
Inclusion Criteria:

* newborn to be operated with the diagnosis of congenital heart disease

Exclusion Criteria:

* age older than 1 month not to be operated

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: This study was conducted in the NICU of Tepecik Training and Research Hospital, İzmir,
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Neutrophil to Lymphocyte Ratio | 1 day
  We measure this with complete blood count to calculate the percentage of neutrophil count to the number of lymphocytes
Neutrophil to Lymphocyte Ratio | 2 week
  We measure this with complete blood count to calculate the percentage of neutrophil count to the number of lymphocytes